CLINICAL TRIAL: NCT05221606
Title: Nurse AMIE (Addressing Malignancies in Individuals Everyday)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH); West Virginia University (Other); Mount Nittany Medical Center (Unknown); Penn State University (Other)
Responsible Party: Principal Investigator, Kathryn Schmitz, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY22090133; R01CA254659 (NIH)
Record Dates: First submitted 2022-01-27; First posted 2022-02-03 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: supportive care; digital health; physical activity; symptom management
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse AMIE Supportive Care Intervention (Experimental): Participants in the intervention arm will receive the computer tablet with the Nurse AMIE program. Nurse AMIE will assess their symptoms daily and provide an intervention to help manage their symptoms.
  Interventions: Behavioral: Nurse AMIE
- Usual Care (Active Comparator): Participants in the usual care arm will receive a book with some supportive care educational materials and recommendations.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Nurse AMIE — Supportive Care Platform (behavioral interventions that are offered based on answers to daily symptom rating questions). Interventions offered include walking, balance, strength exercise, guided relaxation, mindfulness, CBT, DBT, soothing music.
  Arms: Nurse AMIE Supportive Care Intervention
Behavioral: Usual Care — Binder of written supportive care materials
  Arms: Usual Care

SUMMARY:
Nurse AMIE 3.0 is testing the effectiveness of an electronic symptom management system on overall survival in people with stage 3 and 4 cancer who live in rural areas.

DETAILED DESCRIPTION:
After being informed about the details of the study, including risks and potential benefits, participants who give their informed consent will do baseline measurements. After these measures are collected, participants will be randomly assigned to either receive the computer tablet Nurse AMIE program or a supportive care book. Participants will be asked to complete measurements throughout the course of their active participation, which will last for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient receiving care for their cancer
2. Age: 18+ years of age
3. Has stage 3 or 4 cancer, or an unstaged cancer that is considered 'advanced' (greater than stage 2) by their treating oncologist
4. Must be within six months of initiation of pharmacologic or radiation treatment, for curative or palliative purposes, from a medical or radiation oncologist
5. Clinician-rated ECOG function of 0-3
6. Lives in a county with RUCC code 4 - 9 and/or zip code with RUCA code 4-10
7. Has access to personal device capable of receiving telephone calls for study facilitator check-ins
8. Fluent in written and spoken English
9. Sufficient vision/hearing to interact with the tablet and study staff
10. Clinician-defined life expectancy of 6 months or more

Exclusion Criteria:

1. Patients with medical or psychiatric conditions documented in the medical record (beyond cancer, its treatments, and its symptoms) that would impair our ability to test study hypotheses (e.g. psychotic disorders, dementia, inability to give informed consent, or follow study instructions).
2. Patients who are participating in any other supportive care or behavioral intervention studies.
3. Non-English speaking patients will be excluded, as they represent less than 2% of the population targeted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Survival | through study completion, an average of two years
  Survival of each participant will be monitored through the electronic medical records throughout the course of the study. After the study is completed, we will monitor survival using the National Death Index from the Centers for Disease Control and Prevention (CDC).

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life measured using the 36-Item Short Form Health Survey (SF-36) | baseline, month 6, month 12, month 18, month 24
  The SF-36 measures quality of life in the following domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well being, social functioning, pain, and general health. All items are scored from 0 to 100, with 100 being the highest level of functioning possible. Items are averaged to give ratings on each of 8 dimensions.
Change in Physical Function measured using the Short Physical Performance Battery (SPPB) | baseline, month 6, month 12, month 18, month 24
  The SPPB is an accumulation of balance tests, 4-meter gait speed, and 5-chair stands. Based on the time needed to complete the chair stands, a score is given. A summation of scores from all tests is taken, ranging from 0 -12. A higher score = Higher physical function.
Change in Symptoms measured using the Patient-Reported Outcomes Measurement Information System: The PROMIS ®-Preference (PROPr) | baseline, month 1, month 3, month 6, month 9, month 12, month 18, month 24
  The PROMIS PROPr uses 14-items to measure 7 patient symptom domains (two items for each domain). The domains are as follows: cognition, depression, fatigue, pain, physical function, sleep disturbance, and social roles. Scores for each domain range from 1 to 5 on each item, with high scores indicative of full health.
Cost-Effectiveness measured using a self-report survey of Healthcare Utilization | baseline
  This 14-item Healthcare Utilization survey asks participants to account for the healthcare services they used since a key date (provided to the participant). The services include primary care, surgical oncology, medical oncology, other specialists, infusion therapy, radiation therapy, imaging, lab tests, nursing home or rehab stays, hospice, home health care, or other specialty medical care. A high score indicates greater amount of health care services sought.
Cost-Effectiveness measured using a self-report survey of Healthcare Utilization | month1
  This 14-item Healthcare Utilization survey asks participants to account for the healthcare services they used since a key date (provided to the participant). The services include primary care, surgical oncology, medical oncology, other specialists, infusion therapy, radiation therapy, imaging, lab tests, nursing home or rehab stays, hospice, home health care, or other specialty medical care. A high score indicates greater amount of health care services sought.
Cost-Effectiveness measured using a self-report survey of Healthcare Utilization | month 3
  This 14-item Healthcare Utilization survey asks participants to account for the healthcare services they used since a key date (provided to the participant). The services include primary care, surgical oncology, medical oncology, other specialists, infusion therapy, radiation therapy, imaging, lab tests, nursing home or rehab stays, hospice, home health care, or other specialty medical care. A high score indicates greater amount of health care services sought.
Cost-Effectiveness measured using a self-report survey of Healthcare Utilization | month 6
  This 14-item Healthcare Utilization survey asks participants to account for the healthcare services they used since a key date (provided to the participant). The services include primary care, surgical oncology, medical oncology, other specialists, infusion therapy, radiation therapy, imaging, lab tests, nursing home or rehab stays, hospice, home health care, or other specialty medical care. A high score indicates greater amount of health care services sought.
Cost-Effectiveness measured using a self-report survey of Healthcare Utilization | month 9
  This 14-item Healthcare Utilization survey asks participants to account for the healthcare services they used since a key date (provided to the participant). The services include primary care, surgical oncology, medical oncology, other specialists, infusion therapy, radiation therapy, imaging, lab tests, nursing home or rehab stays, hospice, home health care, or other specialty medical care. A high score indicates greater amount of health care services sought.
Cost-Effectiveness measured using a self-report survey of Healthcare Utilization | month 12
  This 14-item Healthcare Utilization survey asks participants to account for the healthcare services they used since a key date (provided to the participant). The services include primary care, surgical oncology, medical oncology, other specialists, infusion therapy, radiation therapy, imaging, lab tests, nursing home or rehab stays, hospice, home health care, or other specialty medical care. A high score indicates greater amount of health care services sought.
Cost-Effectiveness measured using a self-report survey of Healthcare Utilization | month 18
  This 14-item Healthcare Utilization survey asks participants to account for the healthcare services they used since a key date (provided to the participant). The services include primary care, surgical oncology, medical oncology, other specialists, infusion therapy, radiation therapy, imaging, lab tests, nursing home or rehab stays, hospice, home health care, or other specialty medical care. A high score indicates greater amount of health care services sought.
Cost-Effectiveness measured using a self-report survey of Healthcare Utilization | month 24
  This 14-item Healthcare Utilization survey asks participants to account for the healthcare services they used since a key date (provided to the participant). The services include primary care, surgical oncology, medical oncology, other specialists, infusion therapy, radiation therapy, imaging, lab tests, nursing home or rehab stays, hospice, home health care, or other specialty medical care. A high score indicates greater amount of health care services sought.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, Principal Investigator — University of Pittsburgh / UPMC
Locations (8):
- United States (8):
  - UPMC-Butler, Butler, Pennsylvania
  - UPMC - Greenville, Greenville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - UPMC - Indiana, Indiana, Pennsylvania
  - UPMC - New Castle, New Castle, Pennsylvania
  - UPMC - Northwest, Seneca, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmitz KH, Baker S, Werts-Pelter SJ, Doerksen S, Patterson CG, Ahmed M, Scalise R, Vincent A, Desroches C, Sobolewski M, Celebre R, Garrett S, Stout N, Calo WA, Fisher S, Schleicher E, Gordon B, Kumar P. Nurse AMIE randomized controlled trial to address symptom management among rural advanced Cancer patients: Addressing malignancies in everyday life. Contemp Clin Trials. 2025 Aug;155:108005. doi: 10.1016/j.cct.2025.108005. Epub 2025 Jul 10. PMID 40651555

DOCUMENTS (1):
  • Informed Consent Form (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT05221606/ICF_000.pdf